CLINICAL TRIAL: NCT03226873
Title: Assessing the Feasibility and Acceptability of a Peer Outreach and Navigation Intervention to Increase Pre-exposure Prophylaxis Uptake Among Women at High Risk for HIV
Brief Title: Peer Outreach and Navigation Intervention to Increase PrEP Uptake Among Women at High Risk for HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brianna Norton, Assistant Professor of Medicine (GIM), Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-8139; 1U01PS005111-01 (NIH)
Record Dates: First submitted 2017-07-19; First posted 2017-07-24 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Pre-exposure Prophylaxis; HIV-1-infection
Keywords: HIV prevention; PrEP; peer navigation; women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer Navigation (Experimental): PrEP-UP involves a Peer delivering PrEP education and counseling during street-based outreach followed by offer of a PrEP care appointment along with peer navigation (e.g., appointment accompaniment and reminders, etc.) for the first several PrEP visits.
  Interventions: Behavioral: Peer Navigation

INTERVENTIONS:
Behavioral: Peer Navigation — Peer education, counseling, and facilitation of PrEP care

SUMMARY:
This pilot study will assess the feasibility and acceptability of a peer outreach and navigation intervention designed to increase access and promote HIV pre-exposure prophylaxis (PrEP) uptake among women at high risk for HIV.

DETAILED DESCRIPTION:
Women who engage in exchange sex (i.e., sex in exchange for money, drugs, or other services) remain are at substantial risk for HIV infection. (1-6) Due to a confluence of social and structural factors, exchange sex is relatively prevalent among women from socially and economically marginalized groups, such as women who are transgender, unstably housed/homeless and/or those who use and/or inject drugs. (1-3, 19-23) The overarching goal of this research is to decrease new HIV infections among women who engage in exchange sex. Daily oral HIV pre-exposure prophylaxis (PrEP) is an innovative method of HIV prevention that women, themselves, can control; as such, PrEP has the potential to reduce the risk of HIV acquisition among women who engage in exchange sex. Therefore, the investigators developed a theory-guided behavioral intervention (PrEP-UP) which utilizes street-based peer outreach and navigation to increase access to PrEP and promote PrEP uptake among women involved in exchange sex. Specifically, PrEP-UP involves a Peer delivering PrEP education and counseling during street-based outreach followed by offer of a PrEP care appointment along with peer navigation (e.g., appointment accompaniment and reminders, etc.) for the first several PrEP care visits. The objective of this study is to assess the feasibility and acceptability of PrEP-UP. To implement PrEP-UP, the investigators will collaborate with an established community-based organization (CBO) in East Harlem, NY, which uses street-based peer outreach and navigation to connect individuals to needed health and social services. Medical and pharmacy records will be reviewed to assess PrEP initiation. The investigators will conduct self-report surveys at baseline and at a week 4-12 follow-up visit that will collect data about sexual and drug use risk behaviors, perceived HIV risk, and PrEP-related knowledge, attitudes, and self-efficacy to assess for temporal changes in these variables. Additionally, individual interviews will be conducted post-intervention with a subset of the women as well as the CBO staff and leadership to access acceptability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. fluent in English
3. self-identifies as female or male-to-female transgender (or on the spectrum)

Exclusion Criteria

1) Incapable of providing informed consent (i.e., acutely intoxication, active psychosis, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identifying women
Enrollment: 66 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
PrEP prescription filled | 4-12 weeks
  Obtained from medical and/or pharmacy records

SECONDARY OUTCOMES:
HIV risk behaviors | week 0, 4-12
  Revised Risk Behavior Assessment (Wechsberg)
HIV risk perception | week 0, 4-12
  Perceived HIV Risk Scale (Napper)
Interest in PrEP | week 0
  PrEP Acceptability Scale (Marcus)
PrEP appointment acceptance | week 0
  PrEP appointment acceptance (yes/ no)
PrEP appointment scheduled | week 0-12
  Scheduled PrEP appointment (yes/ no)
PrEP appointment attendance | week 0-12
  PrEP appointment attendance (yes/ no)
PrEP-related knowledge | week 0, 4-12
  PrEP Knowledge Scale (Rucinski) (Kalichman) (Kalichman) (Whiteside)
PrEP-related attitudes | week 0, 4-12
  Attitudes Towards PrEP Measurements (Golub) (Holt) (Mimiaga) (Tobias)
PrEP-related self-efficacy | week 0, 4-12
  PrEP Self-Efficacy Scale (adapted from HIV-ASES) (Johnson)

CONTACTS AND LOCATIONS:
Overall Officials: Oni J Blackstock, MD, MHS, Principal Investigator — Albert Einstein College of Medicine; Brianna Norton, DO, MPH, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- New York Harm Reduction Educators, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dunkle KL, Wingood GM, Camp CM, DiClemente RJ. Economically motivated relationships and transactional sex among unmarried African American and white women: results from a U.S. national telephone survey. Public Health Rep. 2010 Jul-Aug;125 Suppl 4(Suppl 4):90-100. doi: 10.1177/00333549101250S413. PMID 20626196
- [Background] Jenness SM, Kobrak P, Wendel T, Neaigus A, Murrill CS, Hagan H. Patterns of exchange sex and HIV infection in high-risk heterosexual men and women. J Urban Health. 2011 Apr;88(2):329-41. doi: 10.1007/s11524-010-9534-5. PMID 21286827
- [Background] Sinoean C. LR, Nerlander L.M., Paz-Bailey G. Prevalence and Correlates of Exchange Sex among Low-Income Heterosexual Women in 21 Cities. Conference on Retroviruses and Opportunistic Infections. Seattle, WA2015.
- [Background] Denning P. HK, Paz-Bailey G.; for the NHBS Study Group. High Levels of HIV Infection Risk among Male Sex Partners of Low-Income Black Women in the United States. International AIDS Society on HIV Pathogenesis. Vancouver, Canada2015.
- [Background] Operario D, Soma T, Underhill K. Sex work and HIV status among transgender women: systematic review and meta-analysis. J Acquir Immune Defic Syndr. 2008 May 1;48(1):97-103. doi: 10.1097/QAI.0b013e31816e3971. PMID 18344875
- [Background] Herbst JH, Jacobs ED, Finlayson TJ, McKleroy VS, Neumann MS, Crepaz N; HIV/AIDS Prevention Research Synthesis Team. Estimating HIV prevalence and risk behaviors of transgender persons in the United States: a systematic review. AIDS Behav. 2008 Jan;12(1):1-17. doi: 10.1007/s10461-007-9299-3. Epub 2007 Aug 13. PMID 17694429
- [Background] Rucinski KB, Mensah NP, Sepkowitz KA, Cutler BH, Sweeney MM, Myers JE. Knowledge and use of pre-exposure prophylaxis among an online sample of young men who have sex with men in New York City. AIDS Behav. 2013 Jul;17(6):2180-4. doi: 10.1007/s10461-013-0443-y. PMID 23479003
- [Background] Kalichman SC, Benotsch E, Suarez T, Catz S, Miller J, Rompa D. Health literacy and health-related knowledge among persons living with HIV/AIDS. Am J Prev Med. 2000 May;18(4):325-31. doi: 10.1016/s0749-3797(00)00121-5. PMID 10788736
- [Background] Kalichman SC, Rompa D. Functional health literacy is associated with health status and health-related knowledge in people living with HIV-AIDS. J Acquir Immune Defic Syndr. 2000 Dec 1;25(4):337-44. doi: 10.1097/00042560-200012010-00007. PMID 11114834
- [Background] Whiteside YO, Harris T, Scanlon C, Clarkson S, Duffus W. Self-perceived risk of HIV infection and attitudes about preexposure prophylaxis among sexually transmitted disease clinic attendees in South Carolina. AIDS Patient Care STDS. 2011 Jun;25(6):365-70. doi: 10.1089/apc.2010.0224. Epub 2011 Apr 6. PMID 21470046
- [Background] Golub SA, Kowalczyk W, Weinberger CL, Parsons JT. Preexposure prophylaxis and predicted condom use among high-risk men who have sex with men. J Acquir Immune Defic Syndr. 2010 Aug;54(5):548-55. doi: 10.1097/QAI.0b013e3181e19a54. PMID 20512046
- [Background] Holt M, Murphy D, Callander D, Ellard J, Rosengarten M, Kippax S, de Wit J. HIV-negative and HIV-positive gay men's attitudes to medicines, HIV treatments and antiretroviral-based prevention. AIDS Behav. 2013 Jul;17(6):2156-61. doi: 10.1007/s10461-012-0313-z. PMID 23001412
- [Background] Mimiaga MJ, Case P, Johnson CV, Safren SA, Mayer KH. Preexposure antiretroviral prophylaxis attitudes in high-risk Boston area men who report having sex with men: limited knowledge and experience but potential for increased utilization after education. J Acquir Immune Defic Syndr. 2009 Jan 1;50(1):77-83. doi: 10.1097/QAI.0b013e31818d5a27. PMID 19295337
- [Background] Tobias CR, Cunningham W, Cabral HD, Cunningham CO, Eldred L, Naar-King S, Bradford J, Sohler NL, Wong MD, Drainoni ML. Living with HIV but without medical care: barriers to engagement. AIDS Patient Care STDS. 2007 Jun;21(6):426-34. doi: 10.1089/apc.2006.0138. PMID 17594252
- [Background] Johnson MO, Neilands TB, Dilworth SE, Morin SF, Remien RH, Chesney MA. The role of self-efficacy in HIV treatment adherence: validation of the HIV Treatment Adherence Self-Efficacy Scale (HIV-ASES). J Behav Med. 2007 Oct;30(5):359-70. doi: 10.1007/s10865-007-9118-3. Epub 2007 Jun 23. PMID 17588200
- [Background] Marcus JL, Glidden DV, Mayer KH, Liu AY, Buchbinder SP, Amico KR, McMahan V, Kallas EG, Montoya-Herrera O, Pilotto J, Grant RM. No evidence of sexual risk compensation in the iPrEx trial of daily oral HIV preexposure prophylaxis. PLoS One. 2013 Dec 18;8(12):e81997. doi: 10.1371/journal.pone.0081997. eCollection 2013. PMID 24367497
- [Background] Wechsberg W. Revised Risk Behavior Assessment (RBA), Part I and Part II. Research Triangle Park, NC: Research Triangle Institute; 1998.
- [Background] Napper LE, Fisher DG, Reynolds GL. Development of the perceived risk of HIV scale. AIDS Behav. 2012 May;16(4):1075-83. doi: 10.1007/s10461-011-0003-2. PMID 21785873
- [Background] Raiford JL, Herbst JH, Carry M, Browne FA, Doherty I, Wechsberg WM. Low prospects and high risk: structural determinants of health associated with sexual risk among young African American women residing in resource-poor communities in the south. Am J Community Psychol. 2014 Dec;54(3-4):243-50. doi: 10.1007/s10464-014-9668-9. PMID 25134798
- [Background] Fletcher JB, Kisler KA, Reback CJ. Housing status and HIV risk behaviors among transgender women in Los Angeles. Arch Sex Behav. 2014 Nov;43(8):1651-61. doi: 10.1007/s10508-014-0368-1. Epub 2014 Sep 5. PMID 25190499
- [Background] Bobashev GV, Zule WA, Osilla KC, Kline TL, Wechsberg WM. Transactional sex among men and women in the south at high risk for HIV and other STIs. J Urban Health. 2009 Jul;86 Suppl 1(Suppl 1):32-47. doi: 10.1007/s11524-009-9368-1. Epub 2009 Jun 10. PMID 19513853
- [Background] Kidder DP, Wolitski RJ, Pals SL, Campsmith ML. Housing status and HIV risk behaviors among homeless and housed persons with HIV. J Acquir Immune Defic Syndr. 2008 Dec 1;49(4):451-5. doi: 10.1097/qai.0b013e31818a652c. PMID 19186357
- [Background] Wechsberg WM, Lam WK, Zule W, Hall G, Middlesteadt R, Edwards J. Violence, homelessness, and HIV risk among crack-using African-American women. Subst Use Misuse. 2003 Feb-May;38(3-6):669-700. doi: 10.1081/ja-120017389. PMID 12747401